CLINICAL TRIAL: NCT01316250
Title: Imatinib Mesylate (Glivec) as Maintenance Therapy After Cytogenetic Response With Nilotinib (AMN107, Tasigna) First Line in Newly Diagnosed Chronic Myelogenous Leukemia
Brief Title: Gleevec as Maintenance Therapy After Cytogenetic Response With Nilotinib in Newly Diagnosed Chronic Myelogenous Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Ali Bazarbachi, Professor, American University of Beirut Medical Center
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: IM.AB.17
Record Dates: First submitted 2011-02-24; First posted 2011-03-16 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: chronic myelogenous leukemia; nilotinib; complete cytogenetic response; imatinib mesylate
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib, cytogenetic response (Other): Newly diagnosed CML patients
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib 300 mg orally twice per day for 12 months followed by imatinib mesylate at a dose of 400 mg orally daily
  Other Names: Tasigna, Gleevec

SUMMARY:
The results of the International Randomized Study of Interferon and STI571 (IRIS) trial indicate that in patients with chronic phase CML treated with first line imatinib, achievement of a complete or partial cytogenetic response (CCyR or PCyR) at 12 months is associated with a significantly better progression-free survival (PFS).

Second generation tyrosine kinase inhibitors such as nilotinib can overcome imatinib resistance because of greater potency to bind to BCR-ABL. Recent results indicate that, in patients with previously untreated chronic phase CML, nilotinib results in a faster and higher rate of CCyR or PCyR than imatinib. However, nilotinib use is associated with diet restriction and much higher financial cost.

The primary objective of this study is to evaluate the ability of imatinib to maintain a complete cytogenetic response (CcyR) in patients who achieved a CCyR after 12 months of first-line treatment with nilotinib.

DETAILED DESCRIPTION:
Imatinib mesylate selectively targets the causative BCR-ABL oncogene in CML. The results of the IRIS trial indicate that in patients with chronic phase CML treated with first line imatinib, achievement of a complete or partial cytogenetic response (CCyR or PCyR) at 12 months is associated with a significantly better progression free survival (PFS).

Second generation tyrosine kinase inhibitors such as nilotinib can overcome imatinib resistance because of greater potency to bind to BCR-ABL. Recent results indicate that, in patients with previously untreated chronic phase CML, nilotinib results in a faster and higher rate of CCyR or PCyR than imatinib. However, nilotinib use is associated with diet restriction and much higher financial cost. Hence, an appealing strategy is to achieve the high rate of CCyR with first line nilotinib and then to maintain this response with long term imatinib which is user friendly and cost-effective.

The primary objective is to test the ability of imatinib to maintain the cytogenetic response in patients who achieved CCyR or PCyR at 12 months with first line nilotinib. The secondary aims are to assess the effects of this strategy on molecular response, BCR-ABL mutations, and CML progenitors.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed untreated Philadelphia chromosome-positive CML (use of hydroxyurea for <3 months is allowed) in chronic phase defined with the following criteria:

   * <15% blasts in peripheral blood (PB) & bone marrow (BM)
   * <30% blasts plus promyelocytes in PB & BM
   * <20% basophils in PB
   * ≥100 x 109/L platelets
   * No evidence of extramedullary involvement, with the exception of liver & spleen
2. Patients (pts) ≥18 yrs of age
3. WHO Performance Status of ≤2
4. Pts must have the following laboratory values:

   * Potassium within normal limits or corrected to within normal limits with supplements prior to the first dose of study medication
   * Total calcium (corrected for serum albumin) and magnesium within normal limits or correctable with supplements
   * Phosphorus ≥ lower limit of normal (LLN) or correctable with supplements
   * ALT and AST ≤2.5 x upper limit of normal (ULN) or ≤5.0xULN if considered due to tumor
   * Alkaline phosphatase ≤2.5xULN
   * Serum bilirubin ≤1.5xULN
   * Serum Cr ≤1.5xULN or 24-hour Cr Cl ≥50 ml/min
   * Serum amylase ≤1.5xULN and serum lipase ≤1.5xULN
5. Written signed informed consent prior to any study procedures

Exclusion Criteria:

1. Cytopathologically confirmed central nervous system (CNS) infiltration
2. Impaired cardiac function, including any one of the following:

   * Left ventricle ejection fraction (LVEF) <45% or below the institutional lower limit of the normal range (whichever is higher) as determined by MUGA scan or echocardiogram
   * Complete left bundle branch block
   * Use of a pacemaker
   * ST depression of >1mm in 2 or more leads and/or T wave inversions in 2 or more contiguous leads
   * Congenital long QT syndrome
   * History of or presence of significant ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia (<50 beats/min)
   * QTc >450 msec on screening ECG
   * Right bundle branch block plus left anterior hemiblock, bifascicular block
   * Myocardial infarction within 12 months prior to starting nilotinib
   * Unstable angina diagnosed or treated during the past 12 months
   * Other clinically significant heart disease (e.g., congestive heart failure, uncontrolled hypertension, or history of labile hypertension)
3. Use of therapeutic coumarin derivatives (i.e., warfarin, acenocoumarol) up to day before study drug administration
4. Acute or chronic liver or renal disease considered unrelated to tumor such as active Hepatitis A, B, or C
5. Other concurrent severe and/or uncontrolled medical conditions
6. Pts who are currently receiving treatment with any of the medications that have the potential to prolong QT interval
7. Pts who have received any investigational drug ≤4 weeks or investigational cytotoxic agent within 1 week (or who are within 5 half-lives of a previous investigational cytotoxic agent) prior to starting study drug or who have not recovered from side effects of such therapy
8. Pts who have received wide field radiotherapy ≤4 weeks or limited field radiation for palliation <2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
9. Pts who have undergone major surgery ≤2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
10. Known diagnosis of HIV
11. Pt with a history of another malignancy that is currently clinically significant or currently requires active intervention
12. Pts who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control (women of childbearing potential must have a negative serum pregnancy test within 48 hrs prior to drug administration). Post menopausal women must be amenorrheic for at least 12 months. Male & female pts must agree to employ an effective method of birth control throughout the study and for 3 months following discontinuation of study drug
13. Pts unwilling or unable to comply with protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2025-07 (Actual); Study Completion 2025-07 (Actual)

PRIMARY OUTCOMES:
To test the ability of imatinib to maintain the cytogenetic response in patients who achieved complete cytogenetic response (CCyR) at 12 months with first line nilotinib. | January 2010-January 2015

SECONDARY OUTCOMES:
To assess the effects of nilotinib followed by imatinib on molecular response | January 2010-January 2015
To assess the effects of nilotinib followed by imatinib on BCR-ABL mutations | January 2010-January 2015

CONTACTS AND LOCATIONS:
Overall Officials: Ali Bazarbachi, MD, PhD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

REFERENCES:
- [Background] Buchdunger E, Cioffi CL, Law N, Stover D, Ohno-Jones S, Druker BJ, Lydon NB. Abl protein-tyrosine kinase inhibitor STI571 inhibits in vitro signal transduction mediated by c-kit and platelet-derived growth factor receptors. J Pharmacol Exp Ther. 2000 Oct;295(1):139-45. PMID 10991971
- [Background] Rosti G, Palandri F, Castagnetti F, Breccia M, Levato L, Gugliotta G, Capucci A, Cedrone M, Fava C, Intermesoli T, Cambrin GR, Stagno F, Tiribelli M, Amabile M, Luatti S, Poerio A, Soverini S, Testoni N, Martinelli G, Alimena G, Pane F, Saglio G, Baccarani M; GIMEMA CML Working Party. Nilotinib for the frontline treatment of Ph(+) chronic myeloid leukemia. Blood. 2009 Dec 3;114(24):4933-8. doi: 10.1182/blood-2009-07-232595. Epub 2009 Oct 12. PMID 19822896
- [Background] Cortes JE, Jones D, O'Brien S, Jabbour E, Konopleva M, Ferrajoli A, Kadia T, Borthakur G, Stigliano D, Shan J, Kantarjian H. Nilotinib as front-line treatment for patients with chronic myeloid leukemia in early chronic phase. J Clin Oncol. 2010 Jan 20;28(3):392-7. doi: 10.1200/JCO.2009.25.4896. Epub 2009 Dec 14. PMID 20008621
- [Background] Druker BJ, Guilhot F, O'Brien SG, Gathmann I, Kantarjian H, Gattermann N, Deininger MW, Silver RT, Goldman JM, Stone RM, Cervantes F, Hochhaus A, Powell BL, Gabrilove JL, Rousselot P, Reiffers J, Cornelissen JJ, Hughes T, Agis H, Fischer T, Verhoef G, Shepherd J, Saglio G, Gratwohl A, Nielsen JL, Radich JP, Simonsson B, Taylor K, Baccarani M, So C, Letvak L, Larson RA; IRIS Investigators. Five-year follow-up of patients receiving imatinib for chronic myeloid leukemia. N Engl J Med. 2006 Dec 7;355(23):2408-17. doi: 10.1056/NEJMoa062867. PMID 17151364
- [Derived] Ibrahim A, Moukalled N, Mahfouz R, El Cheikh J, Bazarbachi A, Abou Dalle I. Safety and Efficacy of Elective Switch from Nilotinib to Imatinib in Newly Diagnosed Chronic Phase Chronic Myeloid Leukemia. Clin Hematol Int. 2022 May 12;4(1-2):30-34. doi: 10.1007/s44228-022-00001-x. eCollection 2022 Jun. PMID 35950205